CLINICAL TRIAL: NCT07170722
Title: Efficacy of Sub-Threshold Dorsal Root Ganglion (DRG) Stimulation Versus Sham in Established Responders: A Randomised, Double-Blind, Two-Period Crossover Trial
Brief Title: Sub-threshold DRG Stimulation vs Sham in Established Responders
Acronym: DRG-SHAM
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Umeå University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Quadruple | Purpose: Treatment
Other Study IDs: DRG-SHAM-2025
Record Dates: First submitted 2025-08-26; First posted 2025-09-12 (Actual); Last update posted 2025-12-05 (Actual); Status verified 2025-08

CONDITIONS: Neuropathic Pain; Complex Regional Pain Syndromes (CRPS); Causalgia; Chronic Pain; Low Back Pain; Pelvic Pain
Keywords: Dorsal Root Ganglion Stimulation; DRG Stimulation; Sub-threshold Stimulation; Neuromodulation; Sham-controlled Trial; Randomized Controlled Trial; Crossover Trial; Chronic Neuropathic Pain; Complex Regional Pain Syndrome (CRPS); Failed Back Surgery Syndrome (FBSS); Post-surgical Pain; Post-traumatic Pain; Low Back Pain; Chronic Pelvic Pain
MeSH Terms: conditions — Neuralgia; Complex Regional Pain Syndromes; Causalgia; Chronic Pain; Low Back Pain; Pelvic Pain; Failed Back Surgery Syndrome; Pain, Postoperative | interventions — salicylhydroxamic acid

STUDY DESIGN:
Intervention Model Description: Randomised, double blinded, sham study
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Subtreshhold DRG-S (Active Comparator): Active Sub-threshold DRG Stimulation Participants receive sub-threshold dorsal root ganglion (DRG) stimulation. Device amplitude is individually titrated to 80% of the perception threshold, ensuring no paresthesia is felt. Frequency and pulse width remain unchanged from each participant's established clinical settings. Stimulation is delivered continuously for 5 days.
  Interventions: Device: Subtreshhold DRG-S
- Sham (Sham Comparator): Sham Stimulation Participants receive sham stimulation. The implanted DRG stimulator is switched off, with device interrogation logs masked to maintain blinding. The sham condition lasts for 5 days.
  Interventions: Other: Sham

INTERVENTIONS:
Device: Subtreshhold DRG-S — Continuous electrical stimulation delivered through an implanted DRG neurostimulator. Amplitude is set individually to 80% of each participant's perception threshold, ensuring no paresthesia is produced. Frequency and pulse width remain unchanged from the participant's established therapeutic settings. This sub-threshold programming distinguishes the intervention from suprathreshold (paresthesia-based) DRG stimulation used in earlier studies.
  Arms: Subtreshhold DRG-S
Other: Sham — The implanted DRG stimulator remains switched off for the entire 5-day period. Device interrogation logs are masked to maintain blinding. No electrical stimulation is delivered, allowing a placebo-controlled comparison with active sub-threshold stimulation.
  Arms: Sham

SUMMARY:
The goal of this clinical trial is to learn if sub-threshold dorsal root ganglion (DRG) stimulation provides pain relief beyond placebo in adults with chronic neuropathic pain who already have an implanted DRG stimulator. The main questions it aims to answer are:

* Does sub-threshold DRG stimulation reduce daily pain intensity compared with sham stimulation?
* How does sub-threshold stimulation affect sleep, mood, and daily activity?

Researchers will compare active sub-threshold DRG stimulation to sham (device switched off) to see if stimulation has a genuine effect on pain and wellbeing.

Participants will:

* Be randomly assigned to receive either active sub-threshold DRG stimulation or sham stimulation for 5 days, followed by the opposite condition for another 5 days.
* Complete short electronic diaries twice daily about their pain, sleep, mood, and activity.
* Attend study visits for safety checks and assessments.

DETAILED DESCRIPTION:
Neuropathic pain is a chronic condition that affects 6-10% of adults and is often resistant to conventional drug therapy. The dorsal root ganglion (DRG) has emerged as an important therapeutic target, as abnormal firing in DRG neurons contributes to peripheral and central sensitization. DRG stimulation (DRGS) delivers mild electrical pulses through implanted leads placed near the DRG. Compared with traditional spinal cord stimulation, DRGS provides highly targeted pain relief with fewer unwanted sensations.

Over the past decade, DRGS has become an established treatment for conditions such as complex regional pain syndrome (CRPS), causalgia, chronic low back pain, and post-surgical neuropathic pain. Modern programming favors sub-threshold settings, in which stimulation is delivered below the level that causes tingling sensations (paresthesias). Although widely adopted, the specific contribution of sub-threshold stimulation has never been confirmed in a sham-controlled trial.

This study is the first randomized, double-blind, sham-controlled trial to directly evaluate whether sub-threshold DRG stimulation provides pain relief beyond placebo. Adults with an implanted DRG stimulator who have shown sustained pain relief will be randomized in a two-period crossover design to receive either active sub-threshold stimulation or sham stimulation, each for 5 days, with a washout period in between.

The primary objective is to determine whether sub-threshold DRG stimulation reduces mean daily pain intensity compared with sham. Secondary objectives include assessing sleep quality, mood, daily activity, and safety/tolerability. Exploratory measures include device logs and rescue medication use.

The findings of this trial will provide critical evidence on the efficacy of sub-threshold DRG stimulation, helping to inform clinical guidelines, payer decisions, and neuromodulation programming strategies worldwide.

ELIGIBILITY:
Inclusion Criteria:

* Adults, age 18 years or older
* Implanted with a dorsal root ganglion (DRG) stimulator for chronic neuropathic pain
* Have experienced at least 50% reduction in pain for 3 months or longer on standard DRG therapy
* Stable pain medication regimen for at least 4 weeks before enrollment
* Able and willing to complete electronic diaries and attend study visits

Exclusion Criteria:

* Active infection or wound complication at the stimulator implant site
* Significant psychiatric illness (for example, uncontrolled depression or psychosis)
* Planned surgery, device reprogramming, or medication changes during the study period
* Currently pregnant or breastfeeding
* Occurrence of any adverse event that meets predefined withdrawal criteria during the study (such as intolerable pain or device-related complications)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2025-09-01 (Actual); Primary Completion 2025-11-30 (Actual); Study Completion 2025-11-30 (Actual)

PRIMARY OUTCOMES:
Average daily pain intensity (Numeric Rating Scale, 0-10) | Twice daily (morning and evening) from Day 0 through Day 11 (includes both 5-day treatment periods and the two 24-hour washout periods on Day 0 and Day 6).
  Self-reported pain intensity recorded twice daily (morning and evening) using an 11-point Numeric Rating Scale (0 = no pain, 10 = worst pain imaginable). Daily scores will be averaged across each treatment and washout period.

SECONDARY OUTCOMES:
Sleep quality (Patient Global Impression of Change, PGIC) | Daily in the morning from Day 0 through Day 11.
  Self-reported sleep quality rated each morning using the Patient Global Impression of Change (PGIC) scale, ranging from 1 = very much worse to 5 = very much improved. Higher scores indicate better sleep.
Mood (Patient Global Impression of Change, PGIC) | Daily in the evening from Day 0 through Day 11.
  Self-reported mood rated each evening using the PGIC scale, ranging from 1 = very much worse to 5 = very much improved. Higher scores indicate better mood.
Daily activity (Patient Global Impression of Change, PGIC) | Daily in the evening from Day 0 through Day 11.
  Self-reported daily activity rated each evening using the PGIC scale, ranging from 1 = very much worse to 5 = very much improved. Higher scores indicate better activity.
Adverse events | From day 0 through end of study (day 11).
  Number and type of adverse events, documented with onset, severity, relatedness to treatment, and resolution.

CONTACTS AND LOCATIONS:
Overall Officials: Pedram Tabatabaei Tabatabaei, M.D, Ph.D, Principal Investigator — Univeristy hospital of northern sweden
Locations (1):
- Neurokirurgiska kliniken. Neuromodulationsenheten, Umeå, Västerbotten County, Sweden

IPD SHARING:
Plan to Share IPD: Yes
De-identified individual participant data (IPD) underlying the published results will be made available. This will include outcome data reported in the manuscript. Data will be available beginning 12 months after publication, with no end date. Access will be granted to qualified researchers upon reasonable request, subject to approval of a proposal and completion of a data use agreement. Data and statistical code will also be deposited in an open repository (OSF)
Supporting Information: Study Protocol, SAP, ICF, CSR
Time Frame: 12 months after publication, with no end date.
Access Criteria: De-identified individual participant data (IPD) underlying the published results, along with the study protocol, statistical analysis plan, and analytic code, will be made available. Access will be provided to qualified researchers affiliated with academic institutions, healthcare organizations, or non-profit entities. Requests must include a research proposal and be approved by the study investigators. Access will be granted under a data use agreement that ensures compliance with GDPR and institutional policies. Data will be hosted in an open-access repository (OSF) 12 months after publication of the primary results.

REFERENCES:
- [Background] Huygen FJPM, Kallewaard JW, Nijhuis H, Liem L, Vesper J, Fahey ME, Blomme B, Morgalla MH, Deer TR, Capobianco RA. Effectiveness and Safety of Dorsal Root Ganglion Stimulation for the Treatment of Chronic Pain: A Pooled Analysis. Neuromodulation. 2020 Feb;23(2):213-221. doi: 10.1111/ner.13074. Epub 2019 Nov 15. PMID 31730273
- [Background] D'Souza RS, Kubrova E, Her YF, Barman RA, Smith BJ, Alvarez GM, West TE, Abd-Elsayed A. Dorsal Root Ganglion Stimulation for Lower Extremity Neuropathic Pain Syndromes: An Evidence-Based Literature Review. Adv Ther. 2022 Oct;39(10):4440-4473. doi: 10.1007/s12325-022-02244-9. Epub 2022 Aug 22. PMID 35994195
- [Background] Deer TR, Levy RM, Kramer J, Poree L, Amirdelfan K, Grigsby E, Staats P, Burton AW, Burgher AH, Obray J, Scowcroft J, Golovac S, Kapural L, Paicius R, Kim C, Pope J, Yearwood T, Samuel S, McRoberts WP, Cassim H, Netherton M, Miller N, Schaufele M, Tavel E, Davis T, Davis K, Johnson L, Mekhail N. Dorsal root ganglion stimulation yielded higher treatment success rate for complex regional pain syndrome and causalgia at 3 and 12 months: a randomized comparative trial. Pain. 2017 Apr;158(4):669-681. doi: 10.1097/j.pain.0000000000000814. PMID 28030470
- [Background] Chapman KB, Sayed D, Lamer T, Hunter C, Weisbein J, Patel KV, Dickerson D, Hagedorn JM, Lee DW, Amirdelfan K, Deer T, Chakravarthy K. Best Practices for Dorsal Root Ganglion Stimulation for Chronic Pain: Guidelines from the American Society of Pain and Neuroscience. J Pain Res. 2023 Mar 14;16:839-879. doi: 10.2147/JPR.S364370. eCollection 2023. PMID 36942306
- [Background] Piedade GS, Gillner S, McPhillips PS, Vesper J, Slotty PJ. Effect of low-frequency dorsal root ganglion stimulation in the treatment of chronic pain. Acta Neurochir (Wien). 2023 Apr;165(4):947-952. doi: 10.1007/s00701-023-05500-1. Epub 2023 Jan 27. PMID 36705762

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2025-09-04): https://cdn.clinicaltrials.gov/large-docs/22/NCT07170722/Prot_SAP_000.pdf